CLINICAL TRIAL: NCT02764450
Title: Marginal Quality of Posterior Microhybrid Resin Composite Restorations Applied Using Two Polymerisation Protocols
Brief Title: 10 Years Evaluation of Composite Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BNM Clinic and Research (Other)
Responsible Party: Principal Investigator, Nicola Barabanti, Principal Investigator, BNM Clinic and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TEX-10y-2016
Record Dates: First submitted 2016-04-08; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Dental Restoration, Permanent
Keywords: composite; restoration; polymerization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astralis 10 HPM (Experimental): Polymerization High-power mode: 1300 mW/cm2 for 10 s
  Interventions: Device: Astralis 10 RM
- Astralis 10 RM (Experimental): Polymerisation regular mode: 650 mW/cm2 for 20
  Interventions: Device: Astralis 10 HPM

INTERVENTIONS:
Device: Astralis 10 HPM — The cavity to be filled is in quadrant I or III
  Arms: Astralis 10 RM
Device: Astralis 10 RM — The cavity to be filled is in quadrant II or IV
  Arms: Astralis 10 HPM

SUMMARY:
This randomised, split-mouth clinical study evaluated the marginal quality of direct Class I and Class II restorations made of microhybrid composite and applied using two polymerisation protocols,

ELIGIBILITY:
Inclusion Criteria:

* subjects at least 18 years old,
* require restorations due to primary caries in contralateral quadrants with opposing and adjacent tooth contact,
* having no restoration in the antagonist,

Exclusion Criteria

* allergic to resin-based materials,
* pregnant or nursing,
* periodontal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2004-04; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of cavity filled with problem in marginal adaptation and in marginal discoloration | 5 years
  Marginal quality of posterior microhybrid resin composite restorations applied using two polymerisation protocols: 5-year randomised split mouth trial.
  The evaluation was done using both SQUACE and USPHS criteria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barabanti N, Gagliani M, Roulet JF, Testori T, Ozcan M, Cerutti A. Marginal quality of posterior microhybrid resin composite restorations applied using two polymerisation protocols: 5-year randomised split mouth trial. J Dent. 2013 May;41(5):436-42. doi: 10.1016/j.jdent.2013.02.009. Epub 2013 Feb 27. PMID 23454329